CLINICAL TRIAL: NCT06311890
Title: Study to Evaluate the Efficacy, Safety and Tolerability of Photodynamic Therapy(PDT) With Chlorin-e6 in Treating Moderate to Severe Acne
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023XLA141-2
Record Dates: First submitted 2024-01-14; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Acne; Photodynamic Therapy
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- photosensitizer group (Experimental): Subjects will receive a photodynamic therapy with chlorin-e6 after acne removal surgery.Each subject will receive three treatments, two weeks (±3 days) intervals.
  Interventions: Drug: N-chlorin e6 triglumine; Procedure: acne removal surgery
- photosensitizer-placebo group (Placebo Comparator): Subjects will receive a red light exposure treatment with chlorin-e6 placebo after acne removal surgery.Each subject will receive three treatments, two weeks (±3 days) intervals.
  Interventions: Procedure: acne removal surgery

INTERVENTIONS:
Drug: N-chlorin e6 triglumine — a photodynamic therapy with chlorin-e6
  Other Names: a red light irradiation
  Arms: photosensitizer group
Procedure: acne removal surgery — acne removal surgery will be given before red light exposure

SUMMARY:
This study aims to evaluate the clinical efficacy, safety and tolerability of a photodynamic therapy(PDT) based on a new photosensitizer, Chlorin-e6, in the treatment of moderate to severe acne. The hypothesis is that the therapy has good efficacy, safety and tolerability.

DETAILED DESCRIPTION:
The acne clinical guidelines all recommend PDT as an alternative therapy for moderate to severe acne based on the excellent performance of ALA-PDT in the treatment of acne vulgaris. Photosensitizers including Porphyrin and Chlorin have also proved to play a positive role in reducing the number of skin lesions and microbial load. Researchers have successfully provided basic evidence that Chlorin-e6 induces inflammation inhibition through AP-1, NF-κB, MAPKs and other pathways of propionibacterium acnes and increases collagen expression in HaCaT cells, which undoubtedly further indicates: As a new type of photosensitive material, Chlorin-e6 derivatives have excellent performance in the face of moderate and severe acne with high levels of inflammation and high risk of scar.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or non-pregnant female 18 years of age and younger than 50 years of age.
2. Subject has moderate to severe facial acne vulgaris.
3. Subject has provided written informed consent.

Exclusion Criteria:

1. People who are taking photosensitive drugs;
2. Allergic to any component of the photosensitizer;
3. porphyrins or allergies to porphyrins, with a history of photosensitivity;
4. Pregnant or lactating women and those planning to become pregnant within 3 months;
5. Oral or topical antibiotics, retinoids, glucocorticoids, peroxybenzoyl and other drugs within the past 1 month;
6. Have a history of exposure to sunlight in the past 1 month, have received photoelectric treatment in the past 3 months, or have received facial grinding treatment in the past six months;
7. are using vasodilators (such as nitroglycerin, etc.), beta blockers (such as metoprolol, etc.), anticoagulants (such as warfarin, etc.) and other drugs that easily cause facial capillary dilatation;
8. Patients with facial rosacea, atopic dermatitis, hormone-dependent dermatitis and other facial skin-related diseases;
9. Abnormal blood and urine routine, liver and kidney function, diseases of important organs and hematopoietic system that researchers believe are not suitable for clinical trials;
10. Patients participating in other clinical trials at the same time.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in Global Acne Grading System (GAGS) Relative to Baseline | Baseline and 2 weeks/1 month/2 month/6 month after final treatment
  The Global Acne Grading System (GAGS) uses the grading score multiplied by the weight of the position, and the cumulative score is 1-18 for mild, 19-30 for moderate, 31-38 for severe, and above 39 for extremely severe.

OTHER OUTCOMES:
Change in Inflammatory&non-inflammatory Lesion Counts Relative to Baseline | Baseline and 2 weeks/1 month/2 month/6 month after final treatment
  Acne, pimple, pustules, and nodules are classified as non-inflammatory and inflammatory in order to evaluate the efficacy of photodynamic anti-inflammatory.
Change in Acne-specific Quality of Life Assessment Instrument（Qol-Acne）Relative to Baseline | Baseline and 2 weeks/1 month/2 month/6 month after final treatment
  Self-perception, social functioning, and emotional functioning were recorded for the most recent week, with a score of 0-3 depending on the choice, with higher scores indicating worse impact of acne on quality of life.
Change in Numerical Rating Scale(NRS) Relative to Baseline | 5 minutes after the start of red light exposure and Immediately after the treatment
  The NRS pain score is the digital pain score, which is used to assess the pain degree of the patient using the Digital Evaluation Scale of Pain Degree. The pain can be divided into different degrees according to the corresponding number, that is, 0 is no pain, 1-3 is mild pain, 4-6 is moderate pain, and 7-10 is severe pain. The higher the score, the higher the pain level and the greater the photodynamic side effects.
Number of participants with abnormalities of Hematological Parameters and Urine Parameters Relative to Baseline | Baseline and 2 weeks after final treatment
  white blood cell count,red blood cell count,haemoglobin,platelet count,ALT,AST,Cr andwhite blood cell count,red blood cell count,Protein in the urine. Clinical Complete blood cell analysis,Liver function,kidney function test and Clinical Urinalysiswill be used as the measurement tools of this result.Normal physiological parameters are regarded as the standard.
  If CREA is higher than normal after PDT or Protein in the urine is higher than normal, renal function may be impaired.If ALT or AST is higher than normal after PDT, liver function may be impaired.If the WBC is higher than normal after PDT, a systemic infection may be present.If RBC or Hb is lower than normal after PDT, anemia may be present.If PLT is lower than normal after PDT, a coagulopathy may be present.If WBC in the urine is higher than normal after PDT, a urinary tract infection may be present.If RBC in the urine is higher than normal after PDT, urological disorders may be present or coagulopathy may be present.
Change in Adverse Reaction Management Form(AR-MF) Relative to Baseline | Baseline and 2 weeks/1 month/2 month/6 month after final treatment
  Adverse Reaction Management Form will be used to systemically investigate the adverse reactions relating to ALA-PDT for acne vulgaris，which including erythema , post-treatment pain, burning skin, dry skin, itching , pustule , edema and blister, or recovery-phase adverse reactions, which included crust, exudation and hyperpigmentation.

CONTACTS AND LOCATIONS:
Overall Officials: Huiyan Chi, doctor, Study Director — Deputy director of dermatology
Locations (1):
- Xiyuan Hospital of China Academy of Chinese Medical Sciences Organization, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 2024.1-2026.9
URL: http://www.xyhospital.com/